CLINICAL TRIAL: NCT01686919
Title: Effect of Milk-free Diet on Weight and Irritable Bowel Syndrome in Morbid Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/966
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Obesity, Morbid
Keywords: Gastric bypass; Questionnaires; Diet; Milk
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- milk-free (Experimental): morbidly obese patients with irritable bowel syndrome (IBS) eligible for gastric bypass surgery
  Interventions: Dietary Supplement: milk-free

INTERVENTIONS:
Dietary Supplement: milk-free — milk-free diet during 8 preoperative weeks

SUMMARY:
Innlandet Hospital in Gjøvik is a center for patients suffering from morbid obesity in Hedmark og Oppland, Norway. Patients with either BMI > 40 kg/m2 or with BMI > 35 kg/m2 and complications who opt for "gastric bypass" surgery, go through a standard program including a thorough clinical examination and information on the operation, followed by a learning and coping program that consists of standard dietary advise for weight loss and includes weekly visits during 8 weeks.

This research project concerns a subgroup in the patient population described above: morbidly obese patients with irritable bowel syndrome (IBS). In this group it will be investigated how an 8 week preoperative milk-free diet affects digestive functions and weight loss. It is known that milk may cause stomach complaints and may make it more difficult to loose weight.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity

Exclusion Criteria:

* no consent
* contraindications to surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
weight loss | 8 weeks

SECONDARY OUTCOMES:
Gastrointestinal symptoms | 8 weeks
  Gastrointestinal symptom rating scale (GSRS-IBS) in validated Norwegian translation
IgG antigen against milk | 8 weeks
  analysed at BMLab, Sandvika

CONTACTS AND LOCATIONS:
Overall Officials: Per Farup, MD prof, Study Director — Norwegian University of Science and Technology